CLINICAL TRIAL: NCT02749682
Title: Impact of Chronic Constipation on the Development Inguinal Hernia
Brief Title: Relationship Between Constipation and Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: Siverek Devlet Hastanesi (Other)
Collaborators: Harran University (Other)
Responsible Party: Principal Investigator, Abdulcabbar Kartal, Principal Investigator, Siverek Devlet Hastanesi
Other Study IDs: 74059997.050.01.04/78
Record Dates: First submitted 2015-10-23; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Inguinal Hernia; Constipation
Keywords: Nyhus classification; constipation severity scale; groin hernia
MeSH Terms: conditions — Hernia, Inguinal; Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- constipation & hernia group: The effect of constipation on study group whether there is a correlation between subgroups of operated patients on the view of direct and indirect hernias(Nyhuss classification).
- constipation & normal population: The level of constipation on normal population using constipation severity scale.

SUMMARY:
The purpose of this study is to asses the effect of chronic constipation on formation of inguinal hernia using Constipation Severity Scale.

DETAILED DESCRIPTION:
Causes of inguinal hernia are known to be multifactorial, although not fully understood. Besides family history, and connective tissue diseases, the sudden increase in abdominal pressure as heavy lifting, chronic constipation , coughing, straining , situations such as difficulty urinating facilitate the formation and emergence of hernia.

Constipation severity scale(CSS) was developed by Varma et al in 2008. CSS is a scale to determine the individuals defecation frequency, the intensity and difficulty during defecation.CSS has three subscales including Pain, Congestion stool and Large Intestine laziness(0-73 points).High scores indicate that serious symptoms.

Investigators found no studies that show how constipation impact on groin hernias. Investigators are planning to understand the effect of constipation on direct and indirect hernia formation.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers(n:100)
* patients above age of 18(n:100)
* patients with groin hernia(n:100)

Exclusion Criteria:

* previous inguinal hernia surgery
* patients who did not accept the procedure
* patients under age of 18

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: study group: 100 patients with groin hernia above age of 18 kontrol group: 100 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Impact of chronic constipation on the development inguinal hernia | 12 months
  This study asses the effect of chronic constipation on formation of inguinal hernia using Constipation Severity Scale(CSS). After the Ethics Committee Approval from Harran University, study was carried out with 200 patient. After filling out a detailed consent form the two groups were asked to fill out the scale(study group: 100 Patients which were operated with the diagnosis of inguinal hernia, control group: 100 volunteers clinically determined to be healthy). . During surgery, hernia types of the patient's in study group defined according to Nyhus classification and noted on the scale. Results in both groups were studied to understand the effect of constipation on development of inguinal hernia and whether there was a correlation between surgical patients and healthy volunteers. The effect of constipation was also evaluated on operated patients on the view of direct and indirect hernias. P <0.05 was considered significant.,

CONTACTS AND LOCATIONS:
Overall Officials: Ali Uzunköy, Study Director — Harran University; Bülent Çitgez, Study Director — Şişli Etfal Hospital

IPD SHARING:
Plan to Share IPD: No